CLINICAL TRIAL: NCT04873024
Title: Real-time Prediction and Prevention of Apnea Events on PAP Machines in an Interventional Study
Brief Title: Prevention of Airway Obstruction Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovaResp Technologies Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional-study
Record Dates: First submitted 2021-04-12; First posted 2021-05-05 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Sleep Apnea, Mixed Central and Obstructive
Keywords: APAP; CPAP; Airway obstructions
MeSH Terms: conditions — Sleep Apnea Syndromes; Airway Obstruction

STUDY DESIGN:
Intervention Model Description: This study has been designed as a single-blind, randomised crossover study, in which recruited patients who suffer from Obstructive Sleep Apnea (OSA) will undergo at least two sleep studies and receive two treatments.
  The intervention arm will be stratified into two groups based on their Obstructive Apnea Index (OAI):
  Group 1 (n=11): Low OAI, 0.8 < OAI < 2.99 and AHI < 5.0 Group 2 (n=11): High OAI, OAI > 3.0, and AHI > 5.0
Who Masked: Participant
Masking Description: Participants will not be informed what treatment will be used during the studies. The device that will be delivering therapy to them will be concealed from view throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-first (Experimental): Participants in this arm will receive the Intervention treatment on the first night, and the control treatment on the second night.
  Interventions: Device: cMAP Flow V 2.0
- Control-first (Experimental): Participants in this arm will receive the Control treatment on the first night, and the Intervention treatment on the second night.
  Interventions: Device: cMAP Flow V 2.0

INTERVENTIONS:
Device: cMAP Flow V 2.0 — Breathing data collected by the device will be processed by a machine learning algorithm to predict obstructive apnea events. When obstructive apnea events are predicted, the algorithm triggers the CPAP device to respond to the apnea event ahead of its onset.
  For the control treatment, the device will operate as its conventional treatment.
  Other Names: Proactive airway management

SUMMARY:
The standard for treatment for people suffering from obstructive sleep apnea (OSA) syndrome involves the use of Continuous, or Automatic Positive Airway Pressure (CPAP, APAP) machines, which work by delivering air via tubing and mask to a patient at pressures of up to 20cmH2O. This increased pressure is meant to stabilize the airway to reduce obstruction events. APAP machines are generally more effective and more comfortable for patients than CPAP machines because these devices automatically adjust pressure to treat an apnea. However, this treatment is reactive and often ineffective since the necessary pressure is applied seconds after breathing has already stopped; The results of a previous study performed showed strong indications for predicting an apnea before it occurs using measurements collected by existing sensors of the CPAP and APAP machines. If apnea events can be predicted before they occur, the air pressure required to treat them could be supplied ahead of time, preventing the apnea from occurring.

The hypothesis to be tested is whether obstructive sleep apnea events can be prevented, by predicting their onset ahead of time and adjusting the airway pressure accordingly.

DETAILED DESCRIPTION:
Patients recruited for the study will undergo two different PAP therapy treatments during sleep: a control treatment and an intervention treatment. Both types of treatment will be delivered using a positive airway pressure (PAP) device with an Investigational Testing Authorization (ITA) from Health Canada (HC). This medical device consists of a commercially available PAP device which has been integrated with a feature to communicate with a computer hosting the predictive software via USB. Using signals received from the PAP device, the software can predict incoming apneas and direct the PAP machine to increase pressure for a short period of time; This study has been designed as a single-blind, randomised crossover study, in which recruited patients who suffer from Obstructive Sleep Apnea (OSA) will undergo at least two sleep studies. During a sleep study, the patient will spend a night of sleep at the sleep clinic (Sleep Disorders Clinic, QEII Abbie J. Lane Memorial Building) and receive one of two PAP therapy treatments; For the control treatment, the PAP device will deliver standard PAP therapy treatment to the patient; For the intervention treatment, the PAP device will deliver the standard PAP therapy treatment in addition to intervention when an apnea is predicted; All recruited participants will undergo at least two study nights and receive both treatments at least once; For all study night, standard Polysomnography (PSG) measurements will also be acquired (breathing rate, brain waves, movement, blood rate, oxygen levels, etc.); Participants will not be told what therapies are being used for each night, and the device used will be concealed from their view; After each night, participants will be asked to fill out a Satisfaction/Adherence questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* No history of self-reported cardiovascular or neurological issues
* Must be a current PAP machine user.
* Must have used PAP machines for more than 4 months.
* Must be at least 18 years old
* Must be able to comply with all study requirements as outlined in the consent form
* Must be able to understand English and be willing to provide written informed consent
* For all nights of the study, participant must be willing to lend their personal PAP device for inspection.
* Must be willing to have their CPAP SD memory card analyzed by OSCAR to determine their average OAI over the past 30 days of use.
* For the low OAI group, participants must have an average OAI between 0.8 - 2.99 and AHI < 5.0 in the past 30 days, which would result in at least one obstructive apnea every two hours each night.
* For the high OAI group, participants must have an average OAI ≥ 3.0 and AHI ≥ 5.0 in the past 30 days, which would result in around 5 obstructive apneas every hour each night.

Exclusion Criteria:

* Subjects actively using bi-level PAP or require oxygen therapy
* History of severe cardiovascular disease, including NYHA Class III or IV heart failure, CAD with angina, or MI/stroke within past 6 months
* Subjects who are medically complicated or who are medically unstable (i.e. cancer, dementia, unstable cardiac or respiratory disease, or unstable psychiatric illness)
* Potential sleep apnea complications that in the opinion of the clinician may affect the health and safety of the participant
* Subjects exhibiting any flu-like or any upper airway tract infection symptoms at the time of assessment
* Pregnant (confirmed verbally)
* Inability or unwillingness of individual to give written informed consent
* Has received bariatric surgery

All participants currently screened, enrolled, and consented who have not yet had all overnight testing done, AND who have an OAI < 3.0 and AHI < 5.0, will be excluded from the study, as this group has been fully enrolled to date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | 2 nights (approx. 8hrs/night)
  To be measured via Polysomnography (PSG) data, which are standard measures obtained in sleep studies. AHI is measured as the average number of Apnea and Hypopnea occurrences in an hour during sleep (units: events/hour).
Obstructive Apnea Index | 2 nights (approx. 8hrs/night)
  To be measured via Polysomnography (PSG) data, which are standard measures obtained in sleep studies. OAI is measured as the average number of exclusively Obstructive Apnea occurrences in an hour during sleep (units: events/hour).
Respiratory Disturbance Index | 2 nights (approx. 8hrs/night)
  To be measured via Polysomnography (PSG) data, which are standard measures obtained in sleep studies.
  RDI is measured as the average number of Apneas, Hypopneas and RERAs (Respiratory Effort Related Arousal) occurrences in an hour during sleep.

SECONDARY OUTCOMES:
Oxygen Desaturation Index (ODI) | 2 nights (approx. 8hrs/night)
  The ODI metric is also obtained through Polysomnography (PSG) data. ODI is measured as the average number of times per hour of sleep that the blood's oxygen level drop by a certain degree from baseline (units: events/hour).
Intervention treatment has an effect on patient adherence | 2 nights (approx. 8hrs/night)
  Another objective will be the comparison of patient satisfaction after each night of sleep, which will be scored and quantified by an adherence/satisfaction questionnaire to determine whether the use of our device had a positive, or neutral effect on their sleep.
  The questionnaire will be given to participants to fill out after treatment.
  Questionnaire responses will be scaled to an Adherence score using a 11-point Likert rating scale. Higher scores indicate higher participant's adherence/satisfaction to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Debra Morrison, M.D., Principal Investigator — Nova Scotia Health
Locations (1):
- Sleep Disorders Clinic, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No